CLINICAL TRIAL: NCT04206397
Title: Mechanisms of Affective Touch in Chronic Pain
Acronym: MATCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laura Case (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Laura Case, Assistant Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 191669; 4R00AT009466-02 (NIH)
Record Dates: First submitted 2019-12-05; First posted 2019-12-20 (Actual); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: affective touch — Various types of touch such as brushing, pressure, and tapping, as well as heat pain

SUMMARY:
This study compares how different types of touch found in massage therapies impact pain perception, and whether these effects differ in individuals with and without chronic pain. This study also examines psychological factors that may predict differences in touch perception in individuals with chronic pain. This research will improve our understanding of whether and how massage therapies can benefit pain and health, and whether this differs in people who suffer from chronic pain.

ELIGIBILITY:
Inclusion Criteria:

1. ages 18-65
2. fluent in English
3. physician diagnosis of Fibromyalgia but no other chronic pain conditions (patients) or no evidence of chronic pain (healthy volunteers)

Exclusion Criteria:

1. Sensory, motor, or anatomic differences or injuries relevant to study procedures
2. Known anomalies of the central nervous system (including stroke, dementia, aneurysm, or personal history of psychosis)
3. Pregnancy
4. Inability to rate pain or sensations
5. Major medical conditions such as kidney, liver, cardiovascular (hypertension, preexisting cardiac arrhythmia), autonomic, pulmonary, or neurological problems (e.g., seizure disorder) or a chronic systemic disease (e.g., diabetes).
6. History of blood clots or first-degree family members with clotting disorders
7. Current use of opiate medication(s)
8. Contraindications to MRI if participating in pilot MRI study
9. Unable to identify a heat stimulus 50C or lower that generates a rating of a 7 on our VAS scale
10. History of fainting or seizures
11. History of frostbite
12. Open cut or sore on hand to be immersed in cold water bath
13. Fracture of limb to be immersed
14. History of Reynaud's phenomenon (hands get white, then blue on exposure to cold, then red on warming)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ACTRI, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fibromyalgia Patients: Adults with diagnosis of Fibromyalgia
- Healthy Controls: Healthy adults with no chronic pain
Period: Overall Study
Arm/Group | Fibromyalgia Patients | Healthy Controls
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fibromyalgia Patients | Healthy Controls | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (14.1) | 39.0 (11.7) | 39.8 (12.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  female | 38 | 37 | 75
  male | 1 | 3 | 4
  other or unknown | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 8 | 20
  Not Hispanic or Latino | 28 | 32 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 9 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 27 | 23 | 50
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Chronic Pain Intensity Using the Chronic Pain Grade Questionnaire
Description: The investigators will measure chronic pain levels using the Characteristic Pain Intensity score, a subscale of the Chronic Pain Grade Questionnaire (CPGQ). The questions that contribute to the subscale each use a scale from 0-10 where 0 is 'no pain' and 10 is 'pain as bad could be', and their mean is multiplied by 10. The intensity subscale score thus ranges from 0 to 100, where 0 would be least pain reported and 100 would be the most pain reported. This measure will be included in a linear regression model to determine whether this measure significantly predicts differences in ratings of touch pleasantness.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fibromyalgia Patients | Healthy Controls
Number analyzed (Participants) | 40 | 40
score on a scale | 66.0 (13.4) | 16.8 (14.2)

2. Primary Outcome: Trauma History Using the Childhood Trauma Questionnaire
Description: The investigators will measure trauma history using the Childhood Trauma Questionnaire. The total score ranges from 25-125, where 25 is the least childhood trauma (better) and 125 is the greatest childhood trauma (worse). This measure will be included in a linear regression model to determine whether this measure significantly predicts differences in ratings of touch pleasantness.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fibromyalgia Patients | Healthy Controls
Number analyzed (Participants) | 40 | 40
score on a scale | 61.6 (10.5) | 55.2 (5.8)

3. Primary Outcome: Current Depression Using the Hospital Anxiety and Depression Scale Without Chronic Pain
Description: The investigators will measure current depression using the Hospital Anxiety and Depression Scale (HADS). The HADS consists of two sub scales for depression and anxiety. The depression sub scale ranges from 0 - 21 where 0 indicates no depression (better) and 21 indicates highest depression levels (worse). This measure will be included in a linear regression model to determine whether this measure significantly predicts differences in ratings of touch pleasantness.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fibromyalgia Patients | Healthy Controls
Number analyzed (Participants) | 40 | 40
score on a scale | 8.2 (4.2) | 3.2 (3.7)

4. Primary Outcome: Ratings of Affective Touch
Description: Touch pleasantness/unpleasantness ratings will be assessed in response to each sensory stimulus (brushing, tapping, and pressure) using a Visual Analog Scale. Anchors were defined as far left = 'extremely unpleasant' (coded as -100), midpoint = 'neutral' (coded as 0), and far right = 'extremely pleasant' (coded as 100). Affective touch perception is defined as the difference in ratings between the affective and neutral touch conditions (rating of brushing minus rating of tapping) during the Day 1 baseline and will be compared between individuals with and without chronic pain. This value ranged from 200 (brushing extremely pleasant and tapping extremely unpleasant) to -200 (tapping extremely pleasant and brushing extremely unpleasant). These values are not inherently 'better' or 'worse' but represent individual differences in preference for affective touch.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fibromyalgia Patients | Healthy Controls
Number analyzed (Participants) | 40 | 40
units on a scale | 18.4 (38.4) | 6.7 (32.2)

5. Primary Outcome: Change in Heat Pain Intensity From Before to After the Cold Water Bath
Description: Pain intensity will be measured before and after the left hand is submerged in cold water (conditioned pain modulation task). Pain intensity will be assessed with a Visual Analog Scale. Anchors are defined as far left = 'no sensation' (coded as -100), midpoint = 'pain threshold' (coded as 0), and far right = 'intolerable pain' (coded as 100). Change in heat pain ratings after cold water bath ranges from -200 to 200 where higher scores indicate pain increases after cold water bath (worse) and lower scores indicate pain reduction (better).
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fibromyalgia Patients | Healthy Controls
Number analyzed (Participants) | 40 | 40
units on a scale | -36.9 (40.3) | -24.3 (28.3)

6. Primary Outcome: Change in Heat Pain Intensity From Before to After Gentle Brushing
Description: Pain intensity will be measured before and after gentle brushing (affective-touch-pain task) on a Visual Analog Scale. Anchors are defined as far left = 'no sensation' (coded as -100), midpoint = 'pain threshold' (coded as 0), and far right = 'intolerable pain' (coded as 100). Change in heat pain ratings after brushing ranges from -200 to 200 where higher scores indicate pain increases (worse) and lower scores indicate pain reduction (better).
Time Frame: Day 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fibromyalgia Patients | Healthy Controls
Number analyzed (Participants) | 40 | 40
units on a scale | -1.2 (25.9) | -7.2 (22.9)

7. Secondary Outcome: Breathing Rate
Description: Respiration rate will be measured during baseline affective touch (brushing).
Time Frame: Day 1
Population: Several participants in each study group were excluded from analysis of breathing rate due to poor quality of respiration recordings, using standardized procedures for data quality review.
Measure: Mean (Standard Deviation); unit: breathes per minute
Arm/Group | Fibromyalgia Patients | Healthy Controls
Number analyzed (Participants) | 35 | 33
breathes per minute | 15.6 (3.9) | 14.7 (3.7)

ADVERSE EVENTS:
Time Frame: Day 1 and Day 2 of the study, plus any contact initiated by the participant to us until study close on October 23, 2024.
Description: Minimal risk study.
Arm/Group | Fibromyalgia Patients | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT04206397/Prot_SAP_001.pdf
  • Informed Consent Form (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT04206397/ICF_000.pdf